CLINICAL TRIAL: NCT06992648
Title: Trifluridine/Tipiracil Plus Regorafenib vs Trifluridine/Tipiracil Plus Bevacizumab for Refractory Metastatic Colorectal Cancer: A Randomized, Controlled, Open-Label, Non-Inferiority Trial
Brief Title: Trifluridine/Tipiracil Plus Regorafenib vs Trifluridine/Tipiracil Plus Bevacizumab for Refractory Metastatic Colorectal Cancer
Acronym: REGTAS-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1454
Record Dates: First submitted 2025-04-15; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Recurrent
Keywords: trifluridine/tipiracil; regorafenib; bevacizumab; non-inferiority; refractory metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil; regorafenib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Trifluridine/tipiracil will be administered orally BID at a starting dose of 30 mg per square meter of body-surface area, on days 1 through 5 every 2 weeks. Regorafenib will be administered orally QD at a dose-escalation strategy (80 mg/day, followed by weekly increase of 40 mg to 120 mg/day), if no significant drug-related adverse events occurred and 120 mg/day for 21 days of a 28-day cycle.
  Interventions: Drug: Trifluridine/Tipiracil + Regorafenib
- Control arm (Active Comparator): Trifluridine/tipiracil will be administered orally BID at a starting dose of 35 mg per square meter of body-surface area, on days 1 through 5 every 2 weeks. Bevacizumab, at a dose of 5 mg per kilogram of body weight, will be administered IV every 2 weeks (day 1 and day 15).
  Interventions: Drug: Trifluridine/tipiracil + bevacizumab

INTERVENTIONS:
Drug: Trifluridine/Tipiracil + Regorafenib — Trifluridine/tipiracil will be administered orally BID at a starting dose of 30 mg per square meter of body-surface area, on days 1 through 5 every 2 weeks. Regorafenib will be administered orally QD at a dose-escalation strategy (80 mg/day, followed by weekly increase of 40 mg to 120 mg/day), if no significant drug-related adverse events occurred and 120 mg/day for 21 days of a 28-day cycle.
  Arms: experimental arm
Drug: Trifluridine/tipiracil + bevacizumab — Trifluridine/tipiracil will be administered orally BID at a starting dose of 35 mg per square meter of body-surface area, on days 1 through 5 every 2 weeks. Bevacizumab, at a dose of 5 mg per kilogram of body weight, will be administered IV every 2 weeks (day 1 and day 15).
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to demonstrate the non-inferiority of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of progression free survival in patients with refractory metastatic colorectal cancer(mCRC) patients. It will also try to estimate the effect of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of OS, ORR, and DCR in patients with refractory mCRC. Other secondary objectives are to compare the safety and tolerance, and the impact on QoL of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in patients with refractory mCRC.

DETAILED DESCRIPTION:
This is an investigator-initiated prospective, multicenter, randomized, controlled, open-label, non-inferiority trial evaluating the efficacy and safety of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in patients with refractory mCRC. The study process consists of:

1. Screening period. After signing the Informed Consent Form (ICF), patients enter the screening period for eligibility assessments. Test results obtained prior to signing the ICF may be used to evaluate inclusion/exclusion criteria if they meet the requirements, and repeat testing is not required after ICF signing.
2. Treatment period. Patients in the experimental arm will receive trifluridine/tipiracil + regorafenib, while those in the control arm will receive trifluridine/tipiracil + bevacizumab. Treatment will continue until the patient experiences disease progression, intolerable toxicity, investigator-determined inability to continue treatment, withdraws the ICF, death or end of study.
3. Follow-up period. After the withdrawal visit, a follow-up will be done every 8 weeks±7 days until death, withdrawal the ICF, loss to follow-up or end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Sign Informed Consent Form (ICF) must be obtained during the screening visit, prior to the performance of any study procedure；
2. Male or female patient aged ≥18 years old;
3. Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded);
4. RAS status must have been previously determined (mutant or wild-type) based on local assessment of tumor biopsy;
5. Prior treatment regimens for the treatment of advanced colorectal cancer must have included a fluoropyrimidine, irinotecan, oxaliplatin, an anti-VEGF monoclonal antibody and/or an anti-EGFR monoclonal antibody for RAS wildtype patients;
6. Has measurable or non-measurable disease as defined by RECIST version 1.1;
7. Is able to swallow oral tablets;
8. Estimated life expectancy ≥12 weeks;
9. ECOG PS 0-1；
10. Has adequate organ function as defined by the following laboratory values obtained within 7 days prior to randomization:

Absolute neutrophil count ≥1.5×109/L; Platelet count ≥75×109/L; Hemoglobin≥90g/L (7 days without transfusion); Creatinine clearance ≥60 mL/min, assessed using the Cockcroft & Gault formula; Total serum bilirubin <1.5×upper limit of normal (ULN) (unless Gilbert disease confirmed); Aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) ≤ 2.5×ULN (unless if liver function abnormalities are due to underlying liver metastasis, AST (SGOT) and ALT (SGPT) ≤ 5×ULN); Urine protein <1+ on urinalysis or 24-hour urine protein <1g; International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN (For patients receiving anti-coagulant therapy the adequate therapeutic levels of PT should be confirmed).

Female of childbearing potential must have been tested negative in a serum pregnancy test within 7 days prior to randomization; All patients must agree to use a highly effective method of birth control as well as their partners during the study and lasting at least 6 months after the last dose.

Exclusion Criteria:

1. Prior trifluridine/tipiracil or TKI regimens for the treatment of advanced colorectal cancer;
2. Pregnancy, lactating female or possibility of becoming pregnant during the study;
3. Patients currently receiving or having received anticancer therapies within 4 weeks prior to randomization;
4. Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy prior to randomization (excluding alopecia, and skin pigmentation);
5. Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease;
6. Has severe or uncontrolled active acute or chronic infection;
7. Has active or history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension;
8. Has any clinically significant active hepatitis, including but not limited to Hepatitis B or Hepatitis C Virus infection;
9. Known carriers of HIV antibodies;
10. Confirmed uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg) or uncontrolled or symptomatic arrhythmia;
11. Deep arterial thromboembolic events including cerebrovascular accident or myocardial infarction within the last 6 months prior to randomization;
12. Major surgery within 4 weeks prior to randomization (the surgical incision should be fully healed prior to study drug administration), or has not recovered from side effects of previous surgery, or patient that may require major surgery during the study;
13. Prior radiotherapy if completed less than 2 weeks before randomization, except if provided as a short course for symptoms palliation only;
14. Other clinically significant medical conditions; Other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 24 months
  The primary objective is to demonstrate the non-inferiority of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of PFS in patients with refractory mCRC

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  To estimate the effect of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of OS in patients with refractory mCRC.
Objective Response Rate（ORR） | up to 36 months
  To estimate the effect of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of ORR in patients with refractory mCRC.
Disease Control Rate（DCR） | up to 36 months
  To estimate the effect of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in terms of DCR in patients with refractory mCRC.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 36 months
  To compare the safety of trifluridine/tipiracil + regorafenib vs trifluridine/tipiracil + bevacizumab in patients with refractory mCRC.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Prof., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Jing Hao, Prof., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No